CLINICAL TRIAL: NCT04472741
Title: Comparison of Newer Colonoscopy Devices With Standard Forward Viewing (SFV) High Definition Colonoscopes in Daily Practice
Brief Title: Comparison of Newer Colonoscopy Devices With Standard Forward Viewing (SFV) Colonoscopes in Daily Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gastroenterologie Baden-Wettingen (Other)
Responsible Party: Principal Investigator, Geyer Martin, Geyer Martin, Director and Principal investigator, Gastroenterologie Baden-Wettingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GastroBaWe
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Adenoma Detection Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FUSE (Other): wide angle colonoscope
  Interventions: Device: difference between colonoscopes
- HD Pentax i10 colonoscopes (Other): SFV instrument
  Interventions: Device: difference between colonoscopes
- Endocuff (Other): Cuff on SFV
  Interventions: Device: difference between colonoscopes

INTERVENTIONS:
Device: difference between colonoscopes — patients have been randomly assigned for colonoscopy with FUSE or HD SFV endoscopes with or without Endocuff

SUMMARY:
Retrospective data analysis of comparsion of 3 types of colonoscopes in daily practice (FUSE Full spectrum colonoscopy with 330° angle of view vs Pentax standard HD-colonoscopes and Pentax plus Endocuff): medical device of the category IIb (CE-marked device used within its intended purpose)

DETAILED DESCRIPTION:
From March 2015 through February 2017 (phase A) patients referred for ambulant colonoscopy in a private Swiss gastroenterologist's practice were alternatingly allocated to one of the two endoscopy theatres. One equipped with a FUSE® endoscopy system from Endochoice (later: Boston Scientific, nA/FUSE®=1044 examinations), the other with an EPKi Processor and Pentax i10 colonoscopes (nA/Pentax=934 examinations). In March 2017 a second doctor joined the practice, but did not contribute to the study. These organizational changes required randomization to be switched from per-patient alternation to per-day alternation in phase B from March 2018 through September 2019. In phase B the FUSE® system was unchanged (nB/FUSE®=1386 examinations), while the Pentax i10 colonoscopes were additionally equipped with Endocuff® (nB/Endocuff®=750 examinations). Patients with contraindica-tion against Endocuff® (known or found diverticular stenosis) were excluded from the study (nB/removed=127). Patients were given their appointments to any free slot throughout the week without stratification. The study and data analysis was consented by the ethical committee EKNZ Ethikkom-mission Nordwest- und Zentralschweiz (Project-ID 2019-01643).

All procedures were performed by one experienced endoscopist (board certified 2004) under nurse assisted propofol sedation (NAPS).

Baseline characteristics, age, sex, BMI, smoking habits, diabetes as well as quality of bowel prepara-tion (measured by BBPS score) and indication for colonoscopy (screening, surveillance, diagnostic, such as diarrhea, bleeding, persistent abdominal pain) were assessed. Amount of sedatives, other medications given during endoscopy (e.g. Buscopan®) and time for the endoscopy e.g. time to ile-um, retraction time (pullback time minus intervention time) and time for intervention were measured by the assistant with a stopwatch. These parameters, polyp counts, size and their localisation (entered in a table and to an anatomical scheme), and satisfaction for all parts of the examination (bowel prep and overall satisfaction) were realtime entered to the database by a tablet computer. The data entry was done coded. Only the main investigator could subdue each single patient.

Statistics were done with a professional statistics, the co-author Dr. Leiner

ELIGIBILITY:
Inclusion Criteria:

* all patient fit for ambulatory colonoscopy

Exclusion Criteria:

* for Endocuff stricturing divertculosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4114 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | within 45 minutes of examination
  adenoma counts

SECONDARY OUTCOMES:
time for endoscopy (time to ileum, withdrawal and intervention time). Medication, Satisfaction on VAS | within 45 minutes of examination
  different endoscopy characteristics

IPD SHARING:
Plan to Share IPD: No